CLINICAL TRIAL: NCT06417788
Title: Dynamic Guided Implant Surgery VS Static Guided Surgery. A Pilot Randomized Clinical Trial.
Brief Title: Dynamic Guided Implant Surgery VS Static Guided Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jordi Marquès Guasch, Jordi marques Guasch, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: CIR-ECL-2018-09
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Partially Edentulous Patients; Bone Crest of at Least 10 mm Length and 6 mm Width; Patients of at Least 18 Years Old
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients who need dental implants and fulfill the inclusion criteria will be randomly allocated to test group (dynamic guided system) or control group (static stereolithographic pilot drill guided system)
Who Masked: Investigator
Masking Description: Due to the nature of the treatment, it is impossible to mask the treatment from the participant and the care provider. However, the data for analysis will be masked to the investigator responsible for assessing the accuracy of each implant placement system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group or Dynamic guided group (Experimental): in this arm, the position and angulation of the implant in the patient's mouth will be guided by a dynamic guided system.
  Interventions: Device: Dental implant placement
- Control group or Static guided group (Active Comparator): In this arm, the position and angulation of the implant in the patient's mouth will be guided by a stereolitographic pilot drill guide.
  Interventions: Procedure: Static guided implant placement

INTERVENTIONS:
Device: Dental implant placement — Dental implant placement guided by Navident® (ClaroNav Inc., Toronto, Canada)
  Other Names: dynamic guided implant placement
  Arms: Test group or Dynamic guided group
Procedure: Static guided implant placement — Dental implant placement guided by a stereolithographic pilot drill guide.
  Other Names: control group
  Arms: Control group or Static guided group

SUMMARY:
This study aims to evaluate if dynamic-guided surgery is an accurate system for placing dental implants.

Researchers will assess the dental implant accuracy of the dynamic guided system compared to the static pilot guide.

Participants will:

* Receive implant treatment that will be placed by a dynamic or static pilot drill guided system.
* Receive post-operative radiological exam for comparative (on the same appointment).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* ASA type 1 or 2,
* Full mouth plaque scores up to 25% (O'LEARY TJ. The plaque control record 1972;43:38), -Partially edentulous with at least one missing tooth
* Having a bone crest of at least 10mm in length and 6mm in width.

Exclusion Criteria:

* medical conditions contraindicating surgery,
* untreated periodontal disease or caries
* the need for bone augmentation
* acute local infections
* history of head/neck radiation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Implant placement accuracy at the implant platform level | The data for the assessment is collected during the same appointment as the implant placement and requires an additional 20 minutes.
  Implant placement accuracy compared with the implant planning. Expressed in mm.
Implant placement accuracy at the implant apex level | The data for the assessment is collected during the same appointment as the implant placement and requires an additional 20 minutes.
  Implant placement accuracy compared with the implant planning. Expressed in mm.
Implant placement accuracy at an angular evel | The data for the assessment is collected during the same appointment as the implant placement and requires an additional 20 minutes.
  Implant placement accuracy compared with the implant planning. Expressed in degrees.
Implant placement accuracy at the vertical plane. | The data for the assessment is collected during the same appointment as the implant placement and requires an additional 20 minutes.
  Implant placement accuracy compared with the implant planning. Expressed in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Plan to publish the IPD.
Supporting Information: SAP, CSR
Time Frame: when the data is available during the publication process

REFERENCES:
- [Background] Somogyi-Ganss E, Holmes HI, Jokstad A. Accuracy of a novel prototype dynamic computer-assisted surgery system. Clin Oral Implants Res. 2015 Aug;26(8):882-890. doi: 10.1111/clr.12414. Epub 2014 May 19. PMID 24837492
- [Background] Van Assche N, Vercruyssen M, Coucke W, Teughels W, Jacobs R, Quirynen M. Accuracy of computer-aided implant placement. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:112-23. doi: 10.1111/j.1600-0501.2012.02552.x. PMID 23062136
- [Background] Hultin M, Svensson KG, Trulsson M. Clinical advantages of computer-guided implant placement: a systematic review. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:124-35. doi: 10.1111/j.1600-0501.2012.02545.x. PMID 23062137
- [Background] Block MS, Emery RW, Lank K, Ryan J. Implant Placement Accuracy Using Dynamic Navigation. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):92-99. doi: 10.11607/jomi.5004. Epub 2016 Sep 19. PMID 27643585
- [Background] D'haese J, Ackhurst J, Wismeijer D, De Bruyn H, Tahmaseb A. Current state of the art of computer-guided implant surgery. Periodontol 2000. 2017 Feb;73(1):121-133. doi: 10.1111/prd.12175. PMID 28000275
- [Background] Sun TM, Lan TH, Pan CY, Lee HE. Dental implant navigation system guide the surgery future. Kaohsiung J Med Sci. 2018 Jan;34(1):56-64. doi: 10.1016/j.kjms.2017.08.011. Epub 2017 Dec 8. PMID 29310817
- [Background] Block MS, Emery RW. Static or Dynamic Navigation for Implant Placement-Choosing the Method of Guidance. J Oral Maxillofac Surg. 2016 Feb;74(2):269-77. doi: 10.1016/j.joms.2015.09.022. Epub 2015 Sep 30. PMID 26452429
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Hendrix JM, Garmon EH. American Society of Anesthesiologists Physical Status Classification System. 2025 Feb 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441940/ PMID 28722969